CLINICAL TRIAL: NCT02511821
Title: Electronic Monitoring of Patient-Reported Outcomes and Function in GI Cancer Surgery: A Feasibility Study
Brief Title: Electronic Monitoring Device of Patient-Reported Outcomes and Function in Improving Patient-Centered Care in Patients With Gastrointestinal Cancer Undergoing Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 15051; NCI-2015-01061 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 15051 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2015-06-26; First posted 2015-07-30 (Estimated); Last update posted 2021-01-07 (Actual); Status verified 2021-01

CONDITIONS: Stage I Adult Liver Cancer; Stage I Colorectal Cancer; Stage IA Gastric Cancer; Stage IA Pancreatic Cancer; Stage IB Gastric Cancer; Stage IB Pancreatic Cancer; Stage II Adult Liver Cancer; Stage IIA Colorectal Cancer; Stage IIA Gastric Cancer; Stage IIA Pancreatic Cancer; Stage IIB Colorectal Cancer; Stage IIB Gastric Cancer; Stage IIB Pancreatic Cancer; Stage IIC Colorectal Cancer; Stage III Pancreatic Cancer; Stage IIIA Adult Liver Cancer; Stage IIIA Colorectal Cancer; Stage IIIA Gastric Cancer; Stage IIIB Adult Liver Cancer; Stage IIIB Colorectal Cancer; Stage IIIB Gastric Cancer; Stage IIIC Adult Liver Cancer; Stage IIIC Colorectal Cancer; Stage IIIC Gastric Cancer; Stage IV Gastric Cancer; Stage IVA Colorectal Cancer; Stage IVA Liver Cancer; Stage IVA Pancreatic Cancer; Stage IVB Colorectal Cancer; Stage IVB Liver Cancer; Stage IVB Pancreatic Cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular; Colorectal Neoplasms; Stomach Neoplasms; Pancreatic Neoplasms; Liver Neoplasms | interventions — Monitoring, Physiologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Supportive Care (Vivofit watch, online surveys) (Experimental): Patients complete online surveys comprising questions about quality of life, symptoms, and activity level, and wear a wristband device (Vivofit watch) 3-7 days prior to and after surgery. After going home, patients complete the symptom survey three times a week and quality of life survey once a week for 2 weeks post-surgery.
  Interventions: Other: Computer-Assisted Intervention; Device: Vivofit watch; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Other: Computer-Assisted Intervention — Complete online surveys
Device: Vivofit watch — Wear Vivofit watch
  Other Names: Monitor
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This pilot clinical trial studies an electronic monitoring device of patient-reported outcomes (PROs) and function in improving patient-centered care in patients with gastrointestinal cancer undergoing surgery. Electronic monitoring is a technology-based way of asking patients about the quality of life, symptoms, and activity using online surveys and an activity tracking watch may make it easier for patients to tell their doctors and nurses about any issues before and after surgery. Electronic systems of assessing PROs may increase the depth and accuracy of available clinical data, save administrative time, prompt early intervention that improves the patient experience, foster patient-provider communication, improve patient safety, and enhance the consistency of data collection across multiple sites.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the feasibility of administration of electronic patient-reported outcomes and functional assessment in gastrointestinal (GI) cancer surgery (gastric, colorectal, liver, pancreas).

II. Determine percentage of patients able to complete > 80% of MD. Anderson Symptom Inventory (MDASI) and European Quality of LIfe-5 Dimensions (EQ-5D) web-based surveys.

III. Determine percentage of patients able to wear the wristband device at least 1 week post-operatively.

IV. Determine length of time to complete the web-based surveys.

V. Determine length of time patients are able to wear the wristband device, before and after surgery.

SECONDARY OBJECTIVES:

I. Determine the percentage of patients who did not enroll in the study and analyze the reasons why. This will be accomplished using: 1) the number of patients asked to participate; 2) the number of patients who declined to participate, and 3) reasons for declining participation.

II. Responses from the Satisfaction Tool will be used to assess: 1) ease of use of web-based surveys and wristband device; 2) feedback on items in the web-based surveys that are distressing or difficult to comprehend; 3) feedback on length of surveys and timing of administration; and 4) suggestions for items that were not covered but should be added.

III. Calculate the mean number of missing items within each questionnaire to identify individual or subsets of questions that are difficult to answer.

OUTLINE:

Patients complete online surveys comprising questions about quality of life, symptoms, and activity level, and wear a wristband device (Vivofit watch) 3-7 days prior to and after surgery. After going home, patients complete the symptom survey three times a week and quality of life survey once a week for 2 weeks post-surgery.

After completion of study, patients are followed up for 1 month.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo surgery for primary or secondary gastric, colorectal, liver, or pancreas cancer
* Able to read and understand English
* Patients across all stages of disease
* There are no restrictions related to performance status or life expectancy
* This protocol is eligible for waiver of informed consent documentation; all subjects must have the ability to understand and the willingness to provide verbal informed consent

Exclusion Criteria:

* Research participants who have no computer and internet access and/or do not use a computer even if one is present in the household
* Subjects, who in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2015-07-22 (Actual); Primary Completion 2016-07-31 (Actual); Study Completion 2016-07-31 (Actual)

PRIMARY OUTCOMES:
Mean time patients are able to tolerate wearing the wristband device, both before and after surgery | Up to 1 month
  Descriptive statistics will be used to describe the distribution of time (before and after surgery) a patient is able to wear the wristband device.
Mean time to complete the web based questionnaires MDASI and EQ-5D, as well as the Self Geriatric Assessment Measure | Up to 1 month
  Descriptive statistics will be used to describe the distribution of time to complete each assessment.
Median time patients are able to tolerate wearing the wristband device, both before and after surgery | Up to 1 month
  Descriptive statistics will be used to describe the distribution of time (before and after surgery) a patient is able to wear the wristband device.
Median time to complete the web based questionnaires MDASI and EQ-5D, as well as the Self Geriatric Assessment Measure | Up to 1 month
  Descriptive statistics will be used to describe the distribution of time to complete each assessment.
Percentage of patients who are able to complete the web-based questionnaires MDASI and EQ-5D | Up to 1 month
  Descriptive statistics will be reported. Patients who complete at least 80% of all scheduled MDASI and EQ-5D questionnaires will be indicated as able to complete the web-based questionnaires. The true population proportion will be estimated with 95% confidence interval of half-width no more than 0.16.
Percentage of patients who are able to wear the wristband device for at least 1 week post-operatively | Up to 1 week post-operatively
  Estimated with 95% confidence interval of half-width no more than 16%.

SECONDARY OUTCOMES:
Ease of use of web-based surveys and wristband device, as measured by responses from Satisfaction Tool | Up to 1 month
Feedback on items in the web-based surveys that are distressing or difficult to comprehend, as measured by responses from Satisfaction Tool | Up to 1 month
Feedback on length of surveys and timing of administration, as measured by responses from Satisfaction Tool | Up to 1 month
Mean number of missing items within each questionnaire | Up to 1 month
  Mean number of missing items within each questionnaire will be calculated to identify individual or subsets of questions that are difficult to answer.
Percentage of patients who did not enroll in the study-composite outcome of multiple measure listed | Up to 1 month
  Percentage of patients who did not enroll in the study will be determined and the reasons why will be analyzed. This will be accomplished using: i) the number of patients asked to participate, ii) the number of patients who declined to participate, and iii) reasons for declining participation.
Suggestions for items that were not covered but should be added, as measured by responses from Satisfaction Tool | Up to 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Virginia Sun, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States